CLINICAL TRIAL: NCT01547143
Title: Pilot Study of First-line Immunosuppressive Therapy Combined With Etoposide and Allogeneic Hematopoietic Cell Transplantation in Refractory/Reactivated Cases for Hemophagocytic Lymphohistiocytosis (HLH) in Adult Patients
Brief Title: Pilot Study of Etoposide-based Therapy and Hematopoietic Cell Transplantation for Hemophagocytic Lymphohistiocytosis
Acronym: HELA2012
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI resigned the institute, and the rest investigators at the institute decided to terminate the study.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-H-72
Record Dates: First submitted 2012-02-29; First posted 2012-03-07 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Secondary hemophagocytic lymphohistiocytosis of adults
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Etoposide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IST and/or alloHCT (Experimental): Patients who are newly diagnosed as HLH by HLH-2004 criteria, excluding those with HLH owing to malignancy or rheumatic disorder.
  Interventions: Drug: IST and/or alloHCT

INTERVENTIONS:
Drug: IST and/or alloHCT — 1) Patients will be categorized by their initial serum ferritin level.
  1. Mild ( ferritin<3,000 μg/L): close observation
  2. Moderate (ferritin: 3,000-10,000 μg/L):
     1. Initiation : cyclosporine 3mg/kg p.o.bid + dexamethasone 10mg/m2/d po. or i.v. (D1-3)
     2. continuation: cyclosporine 3mg/kg p.o. bid (D4-56) + dexamethasone 10mg/m2/d (D4-14), then tapering.
  3. Severe (ferritin>10,000 μg/L):
     1. initiation : etoposide 100mg/m2/d i.v. + cyclosporine 2mg/kg i.v. q 12hours + dexamethasone 20mg/m2/d i.v. (D1-3)
     2. continuation : etoposide 100mg/m2/day weekly (D15-49) + cyclosporine 2mg/kg i.v. q 12 hours? ? po. (D4-56) + dexamethasone 10mg/m2/d (D4-14), 5mg/m2/d (D15-28), 2.5mg/m2/d (D29-42), 1.25mg/m2/d (D43-56), then tapering off.
        2) AlloHCT for refractory or reactivated cases.
  Other Names: Etoposide; Cyclosporine: Cipol; Dexamethasone; IV gammaglobulin

SUMMARY:
The investigators would like to propose a pilot study evaluating the efficacy of etoposide combined with immunosuppressive agents for adult secondary hemophagocytic lymphohistiocytosis (HLH), in order to prove out whether the modification of previous HLH-94 or HLH-2004 protocol for childhood patients can improve the outcome and decrease the toxicities. The results of this pilot study will be a base of a more-improved phase-2 protocol.

DETAILED DESCRIPTION:
The treatment of HLH in adult patients has not been determined yet. Actually, we adopted the treatment protocol HLH2004, which was developed for pediatric HLH patients. The HLH2004 protocol, which is a potent and successful treatment for HLH, has shown some limitations in the treatment of adult HLH. First, the dose of etoposide is somewhat high for adult patients to tolerate. Second, the high incidence of opportunistic infection such as fungal, bacterial, and viral has threatened the patients. Third, more aggressive and intensive approach to adopt allogeneic hematopoietic cell transplantation will be needed earlier in adult patients. Based on these rationales, we developed a modified protocol based on HLH2004 to pit the treatment of adult HLH patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose clinical findings satisfy 5 or more criteria out of the following 8 ones

  1. Fever ≥ 38.5 ℃ for ≥ 7 days
  2. Splenomegaly ≥ 3 FB below left subcostal margin
  3. Cytopenias affecting ≥ 2 of 3 lineages in PB Hb < 9 g/L Platelet < 100 x 109 /L ANC < 1.0 x 109 /L
  4. Hypertriglyceridemia and/or hypofibrinogenemia (fasting triglycerides ≥ 265 mg/dL, fibrinogen ≤ 1.5 g/L)
  5. Hemophagocytosis in BM or spleen or LN
  6. Low or absent NK-cell activity ( according to local laboratory reference)
  7. Serum-ferritin ≥ 500 mcg/L
  8. Soluble CD25(sIL-2 receptor) ≥ 2,400 U/ml
* 18 years of age and over.
* All patients (or his/her family when the patient cannot sign the consent form because of his/her general conditions) give written informed consent according to guidelines at institution's committee on human research.

Exclusion Criteria:

* HLH from malignancy (such as lymphoma, myeloma, leukemia, and other solid tumor)
* HLH from rheumatic disorder (such as SLE, AOSD, antiphospholipid antibody syndrome)
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Male patient who reject the methods of avoiding pregnancy via methods such as abstinence, barrier method (condom etc).
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
overall survival rate | 1-year

SECONDARY OUTCOMES:
Complete response rate | 28 days
Complete response rate | 56 days
Complete response rate | 3 months
Partial response rate | 28 days
Partial response rate | 56 days
Partial response rate | 3 months
reactivation-free survival rate | 3 months
reactivation-free survival rate | 6 months
overall survival rate | 3 months
overall survival rate | 6 months
overall survival rate | 1 year
treatment-related mortality rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Felix FH, Leal LK, Fontenele JB. Cloak and dagger: the case for adult onset still disease and hemophagocytic lymphohistiocytosis. Rheumatol Int. 2009 Jun;29(8):973-4. doi: 10.1007/s00296-008-0825-z. Epub 2008 Dec 30. PMID 19115058
- [Background] Grom AA. Macrophage activation syndrome and reactive hemophagocytic lymphohistiocytosis: the same entities? Curr Opin Rheumatol. 2003 Sep;15(5):587-90. doi: 10.1097/00002281-200309000-00011. PMID 12960485
- [Background] Chen JH, Fleming MD, Pinkus GS, Pinkus JL, Nichols KE, Mo JQ, Perez-Atayde AR. Pathology of the liver in familial hemophagocytic lymphohistiocytosis. Am J Surg Pathol. 2010 Jun;34(6):852-67. doi: 10.1097/PAS.0b013e3181dbbb17. PMID 20442642
- [Background] Ishii E, Ohga S, Imashuku S, Yasukawa M, Tsuda H, Miura I, Yamamoto K, Horiuchi H, Takada K, Ohshima K, Nakamura S, Kinukawa N, Oshimi K, Kawa K. Nationwide survey of hemophagocytic lymphohistiocytosis in Japan. Int J Hematol. 2007 Jul;86(1):58-65. doi: 10.1532/IJH97.07012. PMID 17675268
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360
- [Background] Filipovich AH. Hemophagocytic lymphohistiocytosis (HLH) and related disorders. Hematology Am Soc Hematol Educ Program. 2009:127-31. doi: 10.1182/asheducation-2009.1.127. PMID 20008190
- [Background] Gupta A, Tyrrell P, Valani R, Benseler S, Weitzman S, Abdelhaleem M. The role of the initial bone marrow aspirate in the diagnosis of hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2008 Sep;51(3):402-4. doi: 10.1002/pbc.21564. PMID 18523990
- [Background] Chung HJ, Park CJ, Lim JH, Jang S, Chi HS, Im HJ, Seo JJ. Establishment of a reference interval for natural killer cell activity through flow cytometry and its clinical application in the diagnosis of hemophagocytic lymphohistiocytosis. Int J Lab Hematol. 2010 Apr;32(2):239-47. doi: 10.1111/j.1751-553X.2009.01177.x. Epub 2009 Jul 15. PMID 19614711
- [Background] Allen CE, Yu X, Kozinetz CA, McClain KL. Highly elevated ferritin levels and the diagnosis of hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2008 Jun;50(6):1227-35. doi: 10.1002/pbc.21423. PMID 18085676
- [Background] Lin TF, Ferlic-Stark LL, Allen CE, Kozinetz CA, McClain KL. Rate of decline of ferritin in patients with hemophagocytic lymphohistiocytosis as a prognostic variable for mortality. Pediatr Blood Cancer. 2011 Jan;56(1):154-5. doi: 10.1002/pbc.22774. PMID 20842751
- [Background] Gholam C, Grigoriadou S, Gilmour KC, Gaspar HB. Familial haemophagocytic lymphohistiocytosis: advances in the genetic basis, diagnosis and management. Clin Exp Immunol. 2011 Mar;163(3):271-83. doi: 10.1111/j.1365-2249.2010.04302.x. PMID 21303357
- [Background] Horne A, Ramme KG, Rudd E, Zheng C, Wali Y, al-Lamki Z, Gurgey A, Yalman N, Nordenskjold M, Henter JI. Characterization of PRF1, STX11 and UNC13D genotype-phenotype correlations in familial hemophagocytic lymphohistiocytosis. Br J Haematol. 2008 Oct;143(1):75-83. doi: 10.1111/j.1365-2141.2008.07315.x. Epub 2008 Aug 15. PMID 18710388
- [Background] Marsh RA, Satake N, Biroschak J, Jacobs T, Johnson J, Jordan MB, Bleesing JJ, Filipovich AH, Zhang K. STX11 mutations and clinical phenotypes of familial hemophagocytic lymphohistiocytosis in North America. Pediatr Blood Cancer. 2010 Jul 15;55(1):134-40. doi: 10.1002/pbc.22499. PMID 20486178
- [Background] Meeths M, Entesarian M, Al-Herz W, Chiang SC, Wood SM, Al-Ateeqi W, Almazan F, Boelens JJ, Hasle H, Ifversen M, Lund B, van den Berg JM, Gustafsson B, Hjelmqvist H, Nordenskjold M, Bryceson YT, Henter JI. Spectrum of clinical presentations in familial hemophagocytic lymphohistiocytosis type 5 patients with mutations in STXBP2. Blood. 2010 Oct 14;116(15):2635-43. doi: 10.1182/blood-2010-05-282541. Epub 2010 Jun 17. PMID 20558610
- [Background] Yoon HS, Kim HJ, Yoo KH, Sung KW, Koo HH, Kang HJ, Shin HY, Ahn HS, Kim JY, Lim YT, Bae KW, Lee KO, Shin JS, Lee ST, Chung HS, Kim SH, Park CJ, Chi HS, Im HJ, Seo JJ. UNC13D is the predominant causative gene with recurrent splicing mutations in Korean patients with familial hemophagocytic lymphohistiocytosis. Haematologica. 2010 Apr;95(4):622-6. doi: 10.3324/haematol.2009.016949. Epub 2009 Dec 16. PMID 20015888
- [Background] Arico M, Danesino C, Pende D, Moretta L. Pathogenesis of haemophagocytic lymphohistiocytosis. Br J Haematol. 2001 Sep;114(4):761-9. doi: 10.1046/j.1365-2141.2001.02936.x. No abstract available. PMID 11564062
- [Background] Feldmann J, Callebaut I, Raposo G, Certain S, Bacq D, Dumont C, Lambert N, Ouachee-Chardin M, Chedeville G, Tamary H, Minard-Colin V, Vilmer E, Blanche S, Le Deist F, Fischer A, de Saint Basile G. Munc13-4 is essential for cytolytic granules fusion and is mutated in a form of familial hemophagocytic lymphohistiocytosis (FHL3). Cell. 2003 Nov 14;115(4):461-73. doi: 10.1016/s0092-8674(03)00855-9. PMID 14622600
- [Background] Sieni E, Cetica V, Santoro A, Beutel K, Mastrodicasa E, Meeths M, Ciambotti B, Brugnolo F, zur Stadt U, Pende D, Moretta L, Griffiths GM, Henter JI, Janka G, Arico M. Genotype-phenotype study of familial haemophagocytic lymphohistiocytosis type 3. J Med Genet. 2011 May;48(5):343-52. doi: 10.1136/jmg.2010.085456. Epub 2011 Jan 19. PMID 21248318
- [Background] Chang YH, Lee DS, Jo HS, Cho SI, Yoon HJ, Shin S, Yoon JH, Kim HY, Hong YJ, Hong SI, Cho HI. Tumor necrosis factor alpha promoter polymorphism associated with increased susceptibility to secondary hemophagocytic lymphohistiocytosis in the Korean population. Cytokine. 2006 Oct;36(1-2):45-50. doi: 10.1016/j.cyto.2006.10.010. Epub 2006 Dec 12. PMID 17166738
- [Background] Ishii E, Ueda I, Shirakawa R, Yamamoto K, Horiuchi H, Ohga S, Furuno K, Morimoto A, Imayoshi M, Ogata Y, Zaitsu M, Sako M, Koike K, Sakata A, Takada H, Hara T, Imashuku S, Sasazuki T, Yasukawa M. Genetic subtypes of familial hemophagocytic lymphohistiocytosis: correlations with clinical features and cytotoxic T lymphocyte/natural killer cell functions. Blood. 2005 May 1;105(9):3442-8. doi: 10.1182/blood-2004-08-3296. Epub 2005 Jan 4. PMID 15632205
- [Background] Zhang K, Jordan MB, Marsh RA, Johnson JA, Kissell D, Meller J, Villanueva J, Risma KA, Wei Q, Klein PS, Filipovich AH. Hypomorphic mutations in PRF1, MUNC13-4, and STXBP2 are associated with adult-onset familial HLH. Blood. 2011 Nov 24;118(22):5794-8. doi: 10.1182/blood-2011-07-370148. Epub 2011 Aug 31. PMID 21881043
- [Background] Sumegi J, Barnes MG, Nestheide SV, Molleran-Lee S, Villanueva J, Zhang K, Risma KA, Grom AA, Filipovich AH. Gene expression profiling of peripheral blood mononuclear cells from children with active hemophagocytic lymphohistiocytosis. Blood. 2011 Apr 14;117(15):e151-60. doi: 10.1182/blood-2010-08-300046. Epub 2011 Feb 16. PMID 21325597
- [Background] Imashuku S, Tabata Y, Teramura T, Hibi S. Treatment strategies for Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis (EBV-HLH). Leuk Lymphoma. 2000 Sep;39(1-2):37-49. doi: 10.3109/10428190009053537. PMID 10975382
- [Background] Imashuku S, Kuriyama K, Teramura T, Ishii E, Kinugawa N, Kato M, Sako M, Hibi S. Requirement for etoposide in the treatment of Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis. J Clin Oncol. 2001 May 15;19(10):2665-73. doi: 10.1200/JCO.2001.19.10.2665. PMID 11352958
- [Background] Henter JI, Samuelsson-Horne A, Arico M, Egeler RM, Elinder G, Filipovich AH, Gadner H, Imashuku S, Komp D, Ladisch S, Webb D, Janka G; Histocyte Society. Treatment of hemophagocytic lymphohistiocytosis with HLH-94 immunochemotherapy and bone marrow transplantation. Blood. 2002 Oct 1;100(7):2367-73. doi: 10.1182/blood-2002-01-0172. PMID 12239144
- [Background] Ohga S, Kudo K, Ishii E, Honjo S, Morimoto A, Osugi Y, Sawada A, Inoue M, Tabuchi K, Suzuki N, Ishida Y, Imashuku S, Kato S, Hara T. Hematopoietic stem cell transplantation for familial hemophagocytic lymphohistiocytosis and Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis in Japan. Pediatr Blood Cancer. 2010 Feb;54(2):299-306. doi: 10.1002/pbc.22310. PMID 19827139
- [Background] Cooper N, Rao K, Gilmour K, Hadad L, Adams S, Cale C, Davies G, Webb D, Veys P, Amrolia P. Stem cell transplantation with reduced-intensity conditioning for hemophagocytic lymphohistiocytosis. Blood. 2006 Feb 1;107(3):1233-6. doi: 10.1182/blood-2005-05-1819. Epub 2005 Oct 11. PMID 16219800
- [Background] Marsh RA, Vaughn G, Kim MO, Li D, Jodele S, Joshi S, Mehta PA, Davies SM, Jordan MB, Bleesing JJ, Filipovich AH. Reduced-intensity conditioning significantly improves survival of patients with hemophagocytic lymphohistiocytosis undergoing allogeneic hematopoietic cell transplantation. Blood. 2010 Dec 23;116(26):5824-31. doi: 10.1182/blood-2010-04-282392. Epub 2010 Sep 20. PMID 20855862
- [Background] Durken M, Horstmann M, Bieling P, Erttmann R, Kabisch H, Loliger C, Schneider EM, Hellwege HH, Kruger W, Kroger N, Zander AR, Janka GE. Improved outcome in haemophagocytic lymphohistiocytosis after bone marrow transplantation from related and unrelated donors: a single-centre experience of 12 patients. Br J Haematol. 1999 Sep;106(4):1052-8. doi: 10.1046/j.1365-2141.1999.01625.x. PMID 10520013
- [Background] Jabado N, de Graeff-Meeder ER, Cavazzana-Calvo M, Haddad E, Le Deist F, Benkerrou M, Dufourcq R, Caillat S, Blanche S, Fischer A. Treatment of familial hemophagocytic lymphohistiocytosis with bone marrow transplantation from HLA genetically nonidentical donors. Blood. 1997 Dec 15;90(12):4743-8. PMID 9389690
- [Background] Horne A, Janka G, Maarten Egeler R, Gadner H, Imashuku S, Ladisch S, Locatelli F, Montgomery SM, Webb D, Winiarski J, Filipovich AH, Henter JI; Histiocyte Society. Haematopoietic stem cell transplantation in haemophagocytic lymphohistiocytosis. Br J Haematol. 2005 Jun;129(5):622-30. doi: 10.1111/j.1365-2141.2005.05501.x. PMID 15916685
- [Background] Janka GE. Familial hemophagocytic lymphohistiocytosis. Eur J Pediatr. 1983 Jun-Jul;140(3):221-30. doi: 10.1007/BF00443367. PMID 6354720
- [Background] Cesaro S, Locatelli F, Lanino E, Porta F, Di Maio L, Messina C, Prete A, Ripaldi M, Maximova N, Giorgiani G, Rondelli R, Arico M, Fagioli F. Hematopoietic stem cell transplantation for hemophagocytic lymphohistiocytosis: a retrospective analysis of data from the Italian Association of Pediatric Hematology Oncology (AIEOP). Haematologica. 2008 Nov;93(11):1694-701. doi: 10.3324/haematol.13142. Epub 2008 Sep 2. PMID 18768529
- [Background] Filipovich AH. Hemophagocytic lymphohistiocytosis and related disorders. Curr Opin Allergy Clin Immunol. 2006 Dec;6(6):410-5. doi: 10.1097/01.all.0000246626.57118.d9. PMID 17088644
- [Background] Haddad E, Sulis ML, Jabado N, Blanche S, Fischer A, Tardieu M. Frequency and severity of central nervous system lesions in hemophagocytic lymphohistiocytosis. Blood. 1997 Feb 1;89(3):794-800. PMID 9028310
- [Background] Jordan MB, Filipovich AH. Hematopoietic cell transplantation for hemophagocytic lymphohistiocytosis: a journey of a thousand miles begins with a single (big) step. Bone Marrow Transplant. 2008 Oct;42(7):433-7. doi: 10.1038/bmt.2008.232. Epub 2008 Aug 4. PMID 18679369
- [Background] Imashuku S, Kuriyama K, Sakai R, Nakao Y, Masuda S, Yasuda N, Kawano F, Yakushijin K, Miyagawa A, Nakao T, Teramura T, Tabata Y, Morimoto A, Hibi S. Treatment of Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis (EBV-HLH) in young adults: a report from the HLH study center. Med Pediatr Oncol. 2003 Aug;41(2):103-9. doi: 10.1002/mpo.10314. PMID 12825212
- [Background] Tseng YT, Sheng WH, Lin BH, Lin CW, Wang JT, Chen YC, Chang SC. Causes, clinical symptoms, and outcomes of infectious diseases associated with hemophagocytic lymphohistiocytosis in Taiwanese adults. J Microbiol Immunol Infect. 2011 Jun;44(3):191-7. doi: 10.1016/j.jmii.2011.01.027. Epub 2011 Jan 20. PMID 21524613
- [Background] Park HS, Kim DY, Lee JH, Lee JH, Kim SD, Park YH, Lee JS, Kim BY, Jeon M, Kang YA, Lee YS, Seol M, Lee YJ, Lim YS, Jang S, Park CJ, Chi HS, Lee KH. Clinical features of adult patients with secondary hemophagocytic lymphohistiocytosis from causes other than lymphoma: an analysis of treatment outcome and prognostic factors. Ann Hematol. 2012 Jun;91(6):897-904. doi: 10.1007/s00277-011-1380-3. Epub 2011 Dec 8. PMID 22147006
- [Background] Imashuku S. Treatment of Epstein-Barr virus-related hemophagocytic lymphohistiocytosis (EBV-HLH); update 2010. J Pediatr Hematol Oncol. 2011 Jan;33(1):35-9. doi: 10.1097/MPH.0b013e3181f84a52. PMID 21088619
- [Background] Shin HJ, Chung JS, Lee JJ, Sohn SK, Choi YJ, Kim YK, Yang DH, Kim HJ, Kim JG, Joo YD, Lee WS, Sohn CH, Lee EY, Cho GJ. Treatment outcomes with CHOP chemotherapy in adult patients with hemophagocytic lymphohistiocytosis. J Korean Med Sci. 2008 Jun;23(3):439-44. doi: 10.3346/jkms.2008.23.3.439. PMID 18583880
- [Background] Jin YK, Xie ZD, Yang S, Lu G, Shen KL. Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis: a retrospective study of 78 pediatric cases in mainland of China. Chin Med J (Engl). 2010 Jun;123(11):1426-30. PMID 20819601
- [Background] Raschke RA, Garcia-Orr R. Hemophagocytic lymphohistiocytosis: a potentially underrecognized association with systemic inflammatory response syndrome, severe sepsis, and septic shock in adults. Chest. 2011 Oct;140(4):933-938. doi: 10.1378/chest.11-0619. Epub 2011 Jul 7. PMID 21737492
- [Background] Belyea B, Hinson A, Moran C, Hwang E, Heath J, Barfield R. Spontaneous resolution of Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2010 Oct;55(4):754-6. doi: 10.1002/pbc.22618. PMID 20806367
- [Background] Gupta AA, Tyrrell P, Valani R, Benseler S, Abdelhaleem M, Weitzman S. Experience with hemophagocytic lymphohistiocytosis/macrophage activation syndrome at a single institution. J Pediatr Hematol Oncol. 2009 Feb;31(2):81-4. doi: 10.1097/MPH.0b013e3181923cb4. PMID 19194188
- [Background] Imashuku S, Hibi S, Sako M, Ishida Y, Mugishima H, Chen J, Tsunematsu Y. Soluble interleukin-2 receptor: a useful prognostic factor for patients with hemophagocytic lymphohistiocytosis. Blood. 1995 Dec 15;86(12):4706-7. No abstract available. PMID 8541568
- [Background] Mahlaoui N, Ouachee-Chardin M, de Saint Basile G, Neven B, Picard C, Blanche S, Fischer A. Immunotherapy of familial hemophagocytic lymphohistiocytosis with antithymocyte globulins: a single-center retrospective report of 38 patients. Pediatrics. 2007 Sep;120(3):e622-8. doi: 10.1542/peds.2006-3164. Epub 2007 Aug 14. PMID 17698967